CLINICAL TRIAL: NCT02952248
Title: An Open-label, Phase I Trial to Determine the Maximum-tolerated Dose and Investigate Safety, Pharmacokinetics, and Efficacy of BI 754091 in Patients With Advanced Solid Tumours
Brief Title: A Trial to Find and Investigate a Safe Dose of a New Substance (BI 754091) for Patients With Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1381.1; 2017-005043-33 (EudraCT Number)
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

ARMS (7):
- Phase Ia dose escalation: Cohort 1 (Experimental): Low dose.
  Interventions: Drug: BI 754091
- Phase Ia dose escalation: Cohort 2 (Experimental): Medium dose.
  Interventions: Drug: BI 754091
- Phase Ia dose escalation: Cohort 3 (Experimental): High dose.
  Interventions: Drug: BI 754091
- Phase Ib dose expansion: Cohort 4 (Experimental): Patients with solid tumours including NSCLC, bladder cancer, melanoma, gastric cancer, ovarian cancer, triple-negative breast cancer, and renal-cell cancer
  Interventions: Drug: BI 754091
- Phase Ib dose expansion: Cohort 5 (Experimental): Patients with tumours with high TMB excluding those with high microsatellite instability (MSI-high)
  Interventions: Drug: BI 754091
- Phase Ib dose expansion: Cohort 6 (Experimental): Patients with refractory squamous cell cervical, anal, and skin tumours.
  Interventions: Drug: BI 754091
- Phase Ib dose escalation: Cohort 7 (Experimental): Patients with recurrent human papillomavirus (HPV)-positive, or HPV-negative, vaginal or vulvar squamous cell carcinoma (VSCC)
  Interventions: Drug: BI 754091

INTERVENTIONS:
Drug: BI 754091

SUMMARY:
The main objective of the dose-escalation part of the trial is to determine the safety and tolerability, and to determine the Maximum Tolerated Dose and/or the Recommended Phase 2 Dose (RP2D) of BI 754091 on the basis of patients with dose-limiting toxicities (DLTs) in patients with selected advanced solid malignancies. Safety and tolerability will be evaluated by monitoring the occurrence of adverse events (AEs), serious AEs (SAE), and laboratory parameter abnormalities, as well as changes to vital signs.

Secondary objectives are the determination of the PK profile of BI 754091 after single and multiple doses of BI 754091, and the preliminary assessment of antitumour activity.

In the dose-expansion part of the trial, the main objectives are to further assess the safety, efficacy, PK profile, and biomarkers of BI 754091 in tumours with specific tumour types and/or genetic mutations at the RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written Informed Consent Form (ICF) prior to any trial-specific procedures, sampling, or analyses. If a patient declines to participate in the voluntary pharmacogenetics component of the trial, he/she will not be excluded from other aspects of the trial.
* Patients ≥18 years of age at the time of signature of the ICF
* Phase Ia (dose-escalation)

  * patients with a histologically confirmed diagnosis of advanced, unresectable, and/or metastatic solid tumours (any type).
  * patients who have received all therapy known to confer clinical benefit (including anti-PD-1 or anti-PDL1 therapies, if relevant), or for whom no therapy of proven efficacy exists, or who are not amenable to standard therapies. Patients with anti- PD-1 or anti-PDL1 experience must have a minimum of 60 days between the last dose of the previous anti PD-1/PD-L1 and Cycle 1 Day 1 of BI 754091 treatment.
  * Patients may agree to provide optional paired biopsies.
* Phase Ib (dose expansion)

  * patients with a histologically confirmed diagnosis of select advanced, unresectable, and/or metastatic solid tumours with either 1) high tumor mutation excluding high microsatellite instability or 2) refractory squamous cell cervical, anal and skin tumors, or 3) recurrent vaginal or vulvar squamous cell carcinoma.
  * All patients must have measurable lesions according to Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 must have at least 1 tumour lesion amenable to biopsy, and must be medically fit and willing to undergo a biopsy before first treatment and, unless clinically contraindicated, after 6 weeks on therapy
  * patients who are anti-PD-1 and anti-PDL-1naïve but have failed conventional treatment (excluding anti-PD-1 treatment), or for whom no therapy of proven efficacy exists, or who are not amenable to standard therapies.
* Eastern Cooperative Oncology Group (ECOG) score: 0 to 1
* Life expectancy of at least 12 weeks after the start of the treatment according to the Investigator's judgement
* Females of child-bearing potential willing to use adequate contraceptive measures from the time of screening until 6 months after trial discontinuation, who are not or will not be breast feeding, and agree to have pregnancy tests prior to the start of dosing and at regular visits during the trial. Females not of childbearing potential must have evidence of such by fulfilling one of the following criteria at screening:

  * Post-menopausal: defined as more than 50 years-of-age and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments
  * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy
  * Women under 50 years-of-age would be considered postmenopausal if they have been amenorrhoeic for at least 12 months following the cessation of exogenous hormonal treatments, and have serum follicle-stimulating hormone and luteinizing hormone levels in the postmenopausal range for the institution.
  * For women of childbearing potential using a contraceptive pill, an additional barrier method is necessary. Acceptable highly effective methods of contraception include total sexual abstinence when this is in line with the preferred and usual lifestyle of the study participant (periodic abstinence such as calendar, ovulation, symptothermal, post-ovulation methods and withdrawal are not acceptable methods of contraception), an intrauterine device or intrauterine hormone-releasing system, bilateral tubal ligation, and vasectomised partner (with post-vasectomy proof of absence of sperm)
* Further inclusion criteria apply

Exclusion criteria:

* Major surgery (major according to the Investigator's assessment) performed within 12 weeks prior to first trial treatment or planned within 12 months after screening, e.g.,hip replacement
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial
* Previous enrolment in this trial
* Any investigational or anti-tumour treatment within 4 weeks or 5 half-life period (whichever is shorter) prior to the initial administration of BI 754091.
* Presence of other active invasive cancers other than the one treated in this trial within 5 years prior to screening, with the exception of appropriately treated basal-cell carcinoma of the skin, in situ carcinoma of the uterine cervix, or other local tumours considered cured by local treatment.
* Untreated brain metastasis(es) that may be considered active. Patients with previously treated brain metastases may participate provided they are stable (i.e., without evidence of Progression of Disease by imaging for at least 4 weeks prior to the first dose of trial treatment, and any neurologic symptoms have returned to baseline), and there is no evidence of new or enlarging brain metastases
* Inadequate organ function or bone marrow reserve as demonstrated by the following laboratory values:

  * Absolute neutrophil count <1.5 x 10^9/L (<1500/mm3)
  * Platelet count <100 x 10^9/L
  * Haemoglobin <90 g/L (<9 g/dL)
  * Alanine aminotransferase (ALT) >2.5 times the upper limit of normal (ULN) if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases
  * Aspartate aminotransferase (AST) >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases
  * Total bilirubin >1.5 times ULN, except for patients with Gilbert's syndrome who are excluded if total bilirubin >3.0 x ULN or direct bilirubin >1.5 x ULN
  * Creatinine >1.5 times ULN or creatinine clearance <50 mL/min (measured or calculated by Chronic Kidney Disease Epidemiology (CKD-EPI) Collaboration equation); confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (QTc) >470 msec
  * Any clinically important abnormalities (as assessed by the Investigator) in rhythm, conduction, or morphology of resting Electrocardiograms, e.g., complete left bundle branch block, third degree heart block
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age, or any concomitant medication known to prolong the QT interval
  * Ejection fraction (EF) <55% or the lower limit of normal of the institutional standard will be excluded. Only in cases where the Investigator (or the treating physician or both) suspects cardiac disease with negative effect on the EF will the EF be measured during screening using an appropriate method according to local standards to confirm eligibility (e.g., echocardiogram [ECHO], multi-gated acquisition scan [MUGA]). A historic measurement of EF no older than 6 months prior to first administration of study drug can be accepted provided that there is clinical evidence that the EF value has not worsened since this measurement in the opinion of the Investigator or of the treating physician or both.
* History of pneumonitis within the last 5 years
* History of severe hypersensitivity reactions to other monoclonal Antibodies
* Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of BI 754091
* Active autoimmune disease or a documented history of autoimmune disease, except vitiligo or resolved childhood asthma/atopy
* Known history of human immunodeficiency virus infection or an active hepatitis B or C virus infection. HIV infection is allowed for patients in cohort 6 (cervical/anal squamous) and cohort 7 (vulvar)
* Interstitial lung disease
* Chronic alcohol or drug abuse or any condition that, in the Investigator's opinion, makes him/her an unreliable trial subject, unlikely to complete the trial, or unable to comply with the protocol procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (13):
- United States (7):
  - Florida Cancer Specialists, Sarasota, Florida
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Greenville Health System, Greenville, South Carolina
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Canada (4):
  - Juravinski Cancer Centre - Hamilton Health Sciences, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
- United Kingdom (2):
  - Sarah Cannon Research Institute, London
  - The Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open-label, multicentre, phase 1 trial in patients with advanced solid tumours. Phase Ia dose escalation part consists of 3 cohorts (80, 240 and 400 mg ezabenlimab) to determine the maximum tolerated dose, followed by Phase Ib dose expansion with 4 cohorts to further evaluate safety, pharmacokinetics and efficacy of ezabenlimab.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Phase Ia Dose Escalation: 80 mg Ezabenlimab: 80 milligram (mg) ezabenlimab (BI 754091) solution for infusion after dilution (20mg/mL (vial with 15mL filling volume)) was administered as intravenous infusion on Day 1 of 21-day cycles in patients with advanced solid tumours.
- Phase Ia Dose Escalation: 240 mg Ezabenlimab: 240 milligram (mg) ezabenlimab (BI 754091) solution for infusion after dilution (20mg/mL (vial with 15mL filling volume)) was administered as intravenous infusion on Day 1 of 21-day cycles in patients with advanced solid tumours.
- Phase Ia Dose Escalation: 400 mg Ezabenlimab: 400 milligram (mg) ezabenlimab (BI 754091) solution for infusion after dilution (20mg/mL (vial with 15mL filling volume)) was administered as intravenous infusion on Day 1 of 21-day cycles in patients with advanced solid tumours.
- Phase Ib Dose Expansion: 240 mg Ezabenlimab, 7 Tumours: 240 milligram (mg) ezabenlimab (BI 754091) solution for infusion after dilution (20mg/mL (vial with 15mL filling volume)) was administered as intravenous infusion on Day 1 of 21-day cycles in patients with advanced and/or metastatic solid tumours including non-small cell lung cancer (NSCLC), bladder cancer, melanoma, gastric cancer, ovarian cancer, triple-negative breast cancer (TNBC), and renal cell carcinoma (RCC).
- Phase Ib Dose Expansion: 240 mg Ezabenlimab, High TMB: 240 milligram (mg) ezabenlimab (BI 754091) solution for infusion after dilution (20mg/mL (vial with 15mL filling volume)) was administered as intravenous infusion on Day 1 of 21-day cycles in patients with tumours that are tumour mutational burden (TMB)-high: any tumour with TMBhigh status (>10 mutations/Mb), excluding those that are MSI-high (TMB and MSI status based on any validated test).
- Phase Ib Dose Expansion: 240 mg Ezabenlimab, Cervical/Anal/Skin: 240 milligram (mg) ezabenlimab (BI 754091) solution for infusion after dilution (20mg/mL (vial with 15mL filling volume)) was administered as intravenous infusion on Day 1 of 21-day cycles in patients with squamous cell cervical, anal, and skin tumours that are refractory to standard therapies.
- Phase Ib Dose Expansion: 240 mg Ezabenlimab, VSCC: 240 milligram (mg) ezabenlimab (BI 754091) solution for infusion after dilution (20mg/mL (vial with 15mL filling volume)) was administered as intravenous infusion on Day 1 of 21-day cycles in patients with recurrent human papillomavirus HPV-positive, or HPV-negative, vaginal or vulvar squamous cell carcinoma (VSCC).
Period: Overall Study
Arm/Group | Phase Ia Dose Escalation: 80 mg Ezabenlimab | Phase Ia Dose Escalation: 240 mg Ezabenlimab | Phase Ia Dose Escalation: 400 mg Ezabenlimab | Phase Ib Dose Expansion: 240 mg Ezabenlimab, 7 Tumours | Phase Ib Dose Expansion: 240 mg Ezabenlimab, High TMB | Phase Ib Dose Expansion: 240 mg Ezabenlimab, Cervical/Anal/Skin | Phase Ib Dose Expansion: 240 mg Ezabenlimab, VSCC
Started | 3 | 3 | 3 | 30 | 27 | 31 | 13
Completed | 0 | 0 | 0 | 0 | 3 | 4 | 0
Not Completed | 3 | 3 | 3 | 30 | 24 | 27 | 13
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 3 | 2
Not completed — Progressive disease | 3 | 3 | 3 | 27 | 20 | 22 | 9
Not completed — Missed 2 cycles of treatment due to COVID-19 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Patient decision | 0 | 0 | 0 | 1 | 3 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Clinical progression | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The TS included all participants who received at least 1 dose of ezabenlimab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase Ia Dose Escalation: 80 mg Ezabenlimab | Phase Ia Dose Escalation: 240 mg Ezabenlimab | Phase Ia Dose Escalation: 400 mg Ezabenlimab | Phase Ib Dose Expansion: 240 mg Ezabenlimab, 7 Tumours | Phase Ib Dose Expansion: 240 mg Ezabenlimab, High TMB | Phase Ib Dose Expansion: 240 mg Ezabenlimab, Cervical/Anal/Skin | Phase Ib Dose Expansion: 240 mg Ezabenlimab, VSCC | Total
Number analyzed (Participants) | 3 | 3 | 3 | 30 | 27 | 31 | 13 | 110
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.3 (11.0) | 58.3 (23.8) | 54.7 (7.8) | 64.8 (12.6) | 65.0 (10.7) | 52.5 (13.0) | 63.5 (11.5) | 60.6 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 25 | 16 | 27 | 13 | 84
  Male | 2 | 3 | 1 | 5 | 11 | 4 | 0 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 3 | 2 | 0 | 7
  Not Hispanic or Latino | 3 | 2 | 3 | 29 | 22 | 27 | 13 | 99
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 2 | 5 | 2 | 1 | 11
  White | 2 | 3 | 3 | 25 | 19 | 29 | 12 | 93
  More than one race | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase Ia Dose Escalation: Number of Participants With Dose-limiting Toxicities (DLTs) in the First Cycle (3 Weeks)
Description: Number of participants experiencing dose-limiting toxicities (DLTs) graded according to Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 / 5.0 observed in the first cycle (3 weeks) in order to meet the objective of assessment of the maximum tolerated dose (MTD) of ezabenlimab.
Time Frame: Up to 3 weeks.
Population: Treated Set (TS): The TS included all participants who received at least 1 dose of ezabenlimab. Phase Ia dose escalation.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ia Dose Escalation: 80 mg Ezabenlimab | Phase Ia Dose Escalation: 240 mg Ezabenlimab | Phase Ia Dose Escalation: 400 mg Ezabenlimab
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 0 | 0

2. Primary Outcome: Phase Ib Dose Expansion: Number of Participants With Dose-limiting Toxicities (DLTs) During the Entire Treatment Period
Description: Phase Ib dose expansion: Number of participants with dose-limiting toxicities (DLTs) during the entire treatment period
Time Frame: From first infusion of study treatment until end of study treatment at the time of interim database lock plus 30 days, up to 853 days.
Population: Treated Set (TS): The TS included all participants who received at least 1 dose of ezabenlimab. Phase Ib dose expansion.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib Dose Expansion: 240 mg Ezabenlimab, 7 Tumours | Phase Ib Dose Expansion: 240 mg Ezabenlimab, High TMB | Phase Ib Dose Expansion: 240 mg Ezabenlimab, Cervical/Anal/Skin | Phase Ib Dose Expansion: 240 mg Ezabenlimab, VSCC
Number analyzed (Participants) | 30 | 27 | 31 | 13
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Phase Ib Dose Expansion: Confirmed Objective Response (OR), Defined as the Best Overall Response of Confirmed Complete Response (CR) or Partial Response (PR) According to RECIST v1.1 as Assessed by the Investigator
Description: Confirmed objective Response (OR), defined as the best overall response of confirmed complete response (CR) or partial response (PR) according to RECIST v1.1 assessed by the Investigator, where the best overall response is the best time point response recorded from the first administration of BI 754091 until the earliest of disease progression according to RECIST v1.1, death or last evaluable tumor assessment before start of subsequent anti-cancer therapy, loss to follow- up or withdrawal of consent.
Time Frame: as for outcome 2
Population: Treated Set (TS): The TS included all participants who received at least 1 dose of ezabenlimab. Phase Ib dose expansion. Only participants with post baseline measurements were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib Dose Expansion: 240 mg Ezabenlimab, 7 Tumours | Phase Ib Dose Expansion: 240 mg Ezabenlimab, High TMB | Phase Ib Dose Expansion: 240 mg Ezabenlimab, Cervical/Anal/Skin | Phase Ib Dose Expansion: 240 mg Ezabenlimab, VSCC
Number analyzed (Participants) | 29 | 24 | 31 | 12
Participants | 4 | 4 | 6 | 2

4. Secondary Outcome: Phase Ia Dose Escalation: Confirmed Objective Response According to RECIST v.1.1 as Assessed by the Investigator
Description: Confirmed OR, defined as the best overall response of confirmed complete response (CR) or partial response (PR) according to RECIST v1.1 as assessed by the Investigator where the best overall response is the best time point response recorded from the first administration of BI 754091 until the earliest of disease progression according to RECIST v1.1, death or last evaluable tumor assessment before start of subsequent anti-cancer therapy, loss to follow- up or withdrawal of consent.
Time Frame: From the first administration of BI 754091 until the earliest of disease progression, death or last evaluable tumor assessment before start of subsequent anti-cancer therapy, loss to follow- up or withdrawal of consent, up to 511 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ia Dose Escalation: 80 mg Ezabenlimab | Phase Ia Dose Escalation: 240 mg Ezabenlimab | Phase Ia Dose Escalation: 400 mg Ezabenlimab
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 1 | 0

5. Secondary Outcome: Phase Ia Dose Escalation: Maximum Measured Concentration (Cmax) of Ezabenlimab in Plasma
Description: Maximum measured concentration (Cmax) of ezabenlimab in plasma after single or multiple dose administration of ezabenlimab. Results for cycle 1 and cycle 2 are reported.
Time Frame: 5 minutes prior to BI 754091 infusion start and 0.5, 1, 1.5, 2, 4, 7, 24, 72, 168 and 336 hours after start of BI 754091 infusion.
Population: Pharmacokinetic (PK) analysis set (PKS): The PKS included all patients in the TS who provided at least one evaluable observation for at least one PK endpoint and no PK relevant protocol deviations. Phase Ia dose escalation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram/Milliliter
Arm/Group | Phase Ia Dose Escalation: 80 mg Ezabenlimab | Phase Ia Dose Escalation: 240 mg Ezabenlimab | Phase Ia Dose Escalation: 400 mg Ezabenlimab
Number analyzed (Participants) | 3 | 3 | 3
Microgram/Milliliter
  Cycle 1 | 25.3 (32.7) | 73.7 (9.93) | 128 (27.1)
  Cycle 2 | 33.3 (23.7) | 96.4 (18.3) | 144 (21.9)

6. Secondary Outcome: Phase Ia Dose Escalation: Area Under the Concentration-time Curve of Ezabenlimab in Plasma Over the Time Interval From 0 to 504 Hours (AUC0-504)
Description: Area under the Concentration-time curve of ezabenlimab in plasma over the time interval from 0 to 504 hours (AUC0-504) after single and multiple dose administrations of ezabenlimab. Results for cycle 1 and cycle 2 are reported.
Time Frame: 5 minutes prior to BI 754091 infusion start and 0.5, 1, 1.5, 2, 4, 7, 24, 72, 168, 336 and 504 hours after start of BI 754091 infusion.
Population: Pharmacokinetic (PK) analysis set (PKS): The PKS included all patients in the TS who provided at least one evaluable observation for at least one PK endpoint and no PK relevant protocol deviations. Phase Ia dose escalation. Only participants with non-missing values were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram*hours/milliliter
Arm/Group | Phase Ia Dose Escalation: 80 mg Ezabenlimab | Phase Ia Dose Escalation: 240 mg Ezabenlimab | Phase Ia Dose Escalation: 400 mg Ezabenlimab
Number analyzed (Participants) | 3 | 3 | 3
Microgram*hours/milliliter
  Cycle 1 | 4640 (28.0) | 14300 (19.6) | 22000 (31.9)
  Cycle 2: number analyzed (Participants) | 3 | 2 | 3
  Cycle 2 | 6790 (18.1) | 18800 (21.5) | 28500 (37.1)

7. Secondary Outcome: Phase Ia Dose Escalation: Number of Participants Experiencing Dose-limiting Toxicities (DLTs) From the Start of Treatment Until End of Treatment
Description: Number of participants experiencing dose-limiting toxicities (DLTs), graded according to Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 / 5.0, from the start of treatment until end of treatment (in all cycles) as assessed approximately every 3 weeks.
Time Frame: From first infusion of study treatment until the last infusion of study treatment plus 30 days, up to 511 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ia Dose Escalation: 80 mg Ezabenlimab | Phase Ia Dose Escalation: 240 mg Ezabenlimab | Phase Ia Dose Escalation: 400 mg Ezabenlimab
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 0 | 0

8. Secondary Outcome: Phase Ib Dose Expansion: Confirmed Progression-free Survival (PFS) Defined From Date of Start of Ezabenlimab to the Date of Disease Progression or Death, Whichever Was Earlier, According to RECIST v1.1 as Assessed by the Investigator
Description: Confirmed Progression-free survival (PFS) defined from date of start administration of BI 754091 to the date of disease progression according to RECIST v1.1 as assessed by the Investigator or death from any cause, whichever is earlier.
  PFS according to RECIST v1.1:
  For patients with 'event' as outcome for PFS:
  - PFS [days] = date of outcome - date of first treatment administration + 1
  For patients with 'censored' as outcome for PFS:
  - PFS (censored) [days] = date of outcome - date of first treatment administration+ 1 Median progression free survival time in months is reported.
Time Frame: From first BI 754091 infusion until disease progression or death, whichever is earlier up to 1668 days.
Population: Treated Set (TS): The TS included all participants who received at least 1 dose of ezabenlimab. Phase Ib dose expansion.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Phase Ib Dose Expansion: 240 mg Ezabenlimab, 7 Tumours | Phase Ib Dose Expansion: 240 mg Ezabenlimab, High TMB | Phase Ib Dose Expansion: 240 mg Ezabenlimab, Cervical/Anal/Skin | Phase Ib Dose Expansion: 240 mg Ezabenlimab, VSCC
Number analyzed (Participants) | 30 | 27 | 31 | 13
Months | 1.9 [1.2 to 3.3] | 2.7 [1.3 to NA] — 75th percentile could not be calculated because less than 75% of patients have not reached PFS. | 2.6 [1.4 to 6.1] | 4.2 [1.4 to 5.5]

9. Secondary Outcome: Phase Ib Dose Expansion: Percentage of Participants With Adverse Events (AEs)
Description: Percentage of participants with adverse events (AEs)
Time Frame: From first infusion of study treatment until end of study treatment plus 30 days, up to 1668 days.
Population: Treated Set (TS): The TS included all participants who received at least 1 dose of ezabenlimab. Phase Ib dose expansion.
Measure: Number; unit: Percentage of participants
Arm/Group | Phase Ib Dose Expansion: 240 mg Ezabenlimab, 7 Tumours | Phase Ib Dose Expansion: 240 mg Ezabenlimab, High TMB | Phase Ib Dose Expansion: 240 mg Ezabenlimab, Cervical/Anal/Skin | Phase Ib Dose Expansion: 240 mg Ezabenlimab, VSCC
Number analyzed (Participants) | 30 | 27 | 31 | 13
Percentage of participants | 96.7 | 96.3 | 96.8 | 100.0

10. Secondary Outcome: Phase Ib Dose Expansion: Percentage of Participants With Serious Adverse Events (SAEs)
Description: Percentage of participants with serious adverse events (SAEs).
Time Frame: as for outcome 2
Population: Treated Set (TS): The TS included all participants who received at least 1 dose of ezabenlimab. Phase Ib dose expansion.
Measure: Number; unit: Percentage of participants
Arm/Group | Phase Ib Dose Expansion: 240 mg Ezabenlimab, 7 Tumours | Phase Ib Dose Expansion: 240 mg Ezabenlimab, High TMB | Phase Ib Dose Expansion: 240 mg Ezabenlimab, Cervical/Anal/Skin | Phase Ib Dose Expansion: 240 mg Ezabenlimab, VSCC
Number analyzed (Participants) | 30 | 27 | 31 | 13
Percentage of participants | 33.3 | 25.9 | 48.4 | 46.2

11. Secondary Outcome: Phase Ib Dose Expansion: Percentage of Participants With Clinically Relevant Abnormalities in Laboratory Evaluations
Description: Percentage of participants with clinically relevant abnormalities in laboratory evaluations is reported by the percentage of participants with liver enzyme elevations.
  Abbreviations:
  ALT: Alanine aminotransferase ALP: Alkaline Phosphatase AST: Aspartate aminotransferase ULN: Upper limit of normal
  *: Tbili elevation must be within +/- 30 days of ALT and/or AST elevation
Time Frame: From first infusion of study treatment until end of study treatment plus 30 days, up to 1668 days.
Population: Treated Set (TS): The TS included all participants who received at least 1 dose of ezabenlimab. Phase Ib dose expansion.
Measure: Number; unit: Percentage of participants
Arm/Group | Phase Ib Dose Expansion: 240 mg Ezabenlimab, 7 Tumours | Phase Ib Dose Expansion: 240 mg Ezabenlimab, High TMB | Phase Ib Dose Expansion: 240 mg Ezabenlimab, Cervical/Anal/Skin | Phase Ib Dose Expansion: 240 mg Ezabenlimab, VSCC
Number analyzed (Participants) | 30 | 27 | 31 | 13
Percentage of participants
  Maximum ALT; >= 3x ULN and <5x ULN | 3.3 | 3.7 | 0.0 | 0.0
  Maximum AST; >= 3x ULN and <5x ULN | 0.0 | 11.1 | 0.0 | 7.7
  Maximum AST; >= 5x ULN and <10x ULN | 3.3 | 0.0 | 0.0 | 0.0
  Maximum Total Bilirubin; >=2x ULN | 0.0 | 11.1 | 3.2 | 0.0
  ALT and/or AST >= 3xULN and * total bilirubin >= 2xULN | 0.0 | 3.7 | 0.0 | 0.0
  Maximum ALP; >=3x ULN and <5x ULN | 3.3 | 11.1 | 3.2 | 0.0
  Maximum ALP; >=5x ULN and <10x ULN | 0.0 | 14.8 | 3.2 | 0.0

ADVERSE EVENTS:
Time Frame: All-cause Mortality: From study start until end of study, up to 2444 days. Serious and other AEs: From treatment start until end of treatment, plus 30 days of residual effect period, up to 511 days for phase Ia dose escalation and up to 1668 days for phase Ib dose expansion.
Description: Treated Set (TS): The TS included all patients who received at least 1 dose of ezabenlimab.
Arm/Group | Phase Ia Dose Escalation: 80 mg Ezabenlimab | Phase Ia Dose Escalation: 240 mg Ezabenlimab | Phase Ia Dose Escalation: 400 mg Ezabenlimab | Phase Ib Dose Expansion: 240 mg Ezabenlimab, 7 Tumours | Phase Ib Dose Expansion: 240 mg Ezabenlimab, High TMB | Phase Ib Dose Expansion: 240 mg Ezabenlimab, Cervical/Anal/Skin | Phase Ib Dose Expansion: 240 mg Ezabenlimab, VSCC
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 2/3 | 16/30 | 10/27 | 17/31 | 9/13
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 2/3 | 10/30 | 9/27 | 16/31 | 6/13
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 27/30 | 24/27 | 30/31 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ia Dose Escalation: 80 mg Ezabenlimab (N=3) | Phase Ia Dose Escalation: 240 mg Ezabenlimab (N=3) | Phase Ia Dose Escalation: 400 mg Ezabenlimab (N=3) | Phase Ib Dose Expansion: 240 mg Ezabenlimab, 7 Tumours (N=30) | Phase Ib Dose Expansion: 240 mg Ezabenlimab, High TMB (N=27) | Phase Ib Dose Expansion: 240 mg Ezabenlimab, Cervical/Anal/Skin (N=31) | Phase Ib Dose Expansion: 240 mg Ezabenlimab, VSCC (N=13)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Biliary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 3 | 0
Spontaneous bacterial peritonitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Urogenital fistula (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Foot amputation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Embolism venous (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ia Dose Escalation: 80 mg Ezabenlimab (N=3) | Phase Ia Dose Escalation: 240 mg Ezabenlimab (N=3) | Phase Ia Dose Escalation: 400 mg Ezabenlimab (N=3) | Phase Ib Dose Expansion: 240 mg Ezabenlimab, 7 Tumours (N=30) | Phase Ib Dose Expansion: 240 mg Ezabenlimab, High TMB (N=27) | Phase Ib Dose Expansion: 240 mg Ezabenlimab, Cervical/Anal/Skin (N=31) | Phase Ib Dose Expansion: 240 mg Ezabenlimab, VSCC (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 9 | 7 | 5
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 3
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 4 | 3 | 4 | 2
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Swelling of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 2 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 5 | 5 | 5 | 1
Chapped lips (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 4 | 3 | 6 | 5
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 5 | 5 | 5 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 3 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 9 | 5 | 9 | 8
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal tenesmus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 6 | 4 | 2
Asthenia (General disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 2 | 1 | 2 | 1
Chills (General disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 2
Fatigue (General disorders) | 1 | 1 | 2 | 12 | 6 | 16 | 5
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0 | 3 | 3 | 8 | 3
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1 | 1 | 4 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 3 | 1 | 6 | 3
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Nail bed infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 3 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 2 | 9 | 4
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Vulvitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 3
Blood creatine increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 2 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 2 | 2 | 2 | 5 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2 | 6 | 5 | 6 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 2 | 4 | 5 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 3 | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 5 | 2 | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 7 | 2 | 5 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5 | 2 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 3 | 3 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 3 | 4 | 4
Pubic pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 3 | 1 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 4 | 3 | 3 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0 | 1 | 7 | 2
Mental fatigue (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1
Vaginal odour (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vulval disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulval ulceration (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Vulvovaginal swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 6 | 1 | 8 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 7 | 1 | 5 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 2 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 3 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 1
Itching scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 4 | 3 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3 | 3 | 4 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3 | 2 | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cataract operation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0
Peripheral vein stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT02952248/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT02952248/SAP_001.pdf